CLINICAL TRIAL: NCT03628781
Title: Improving ADHD Behavioral Care Quality in Community-Based Pediatric Settings
Brief Title: Improving ADHD Behavioral Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeff Epstein, Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18HS024690 (AHRQ)
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Results first posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2021-12

CONDITIONS: ADHD
Keywords: Behavioral intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mehealth portal with integrated behavioral tools (Experimental): Patients in this arm will continue to use the mehealth for ADHD web-based software for ADHD care but will also have access to a module that allows parents and teachers to develop and implement behavioral interventions such as daily report cards online.
  Interventions: Other: Behavioral tools integrated within mehealth for ADHD software; Other: mehealth for ADHD
- mehealth portal with no integrated behavioral tools (Other): Patients in this arm will continue to use the mehealth for ADHD web-based software for ADHD care but will wait one year before getting access to the behavioral intervention features.
  Interventions: Other: mehealth for ADHD

INTERVENTIONS:
Other: Behavioral tools integrated within mehealth for ADHD software — Integrated functionality within the mehealth for ADHD software allows parents and teachers to set up and deliver behavioral interventions such as daily report card systems and home-based program such as star charts. Automated wizards lead parents and teachers through the process of selecting target behaviors and setting up reward schedules. Baseline data is gathered online and algorithms derive a set of behavioral goals for the child. Thereafter, parents or teachers record the child's performance directly into the software. Once behavioral monitoring begins, parents and teachers receive daily email or text communications from mehealth for ADHD alerting them to the daily rewards earned by their child. Finally, online algorithms exist that detect how a child is doing in meeting behavioral goals and prompt users to modify goals accordingly.
  Arms: mehealth portal with integrated behavioral tools
Other: mehealth for ADHD — The mehealth for ADHD software has multiple functionalities including 1) online training regarding the American Academy of Pediatrics (AAP) ADHD guidelines; 2) an ADHD workflow wizard that guides pediatricians through the creation of an efficient office workflow to deliver quality ADHD care; 3) online collection of parent- and teacher-report ADHD rating scales for the assessment of ADHD as well as monitoring response to medication treatment; 4) integrated algorithms that automatically score rating scales in real time and provide pediatricians with assessment and treatment reports as well as immediate warnings; 5) a communication feature that allows parents, teachers, and pediatricians to communicate with each other; 6) an online pediatrician "report card"; and 7) a Plan-Do-Study-Act wizard that allows pediatricians to select a practice behavior to improve based on their report card and guides them through the creation of small tests of change to improve their office systems.

SUMMARY:
Though the most effective treatment for children with Attention Deficit Hyperactivity Disorder (ADHD) consists of combined medication and behavioral strategies, the vast majority of children with ADHD are treated with medication only. One reason for the low rates of behavioral treatment is that primary care pediatricians, not mental health professionals, are responsible for treating the vast majority of children with ADHD. The investigators have developed, tested, and are beginning to disseminate web-based software (mehealth for ADHD) that has been shown in randomized clinical trials to improve the quality of ADHD medication care delivered by pediatricians. The goal of the proposed study is to develop and test the integration of behavioral tools into the evidence-based myadhdportal.com software in order to improve access to behavioral treatment strategies, and ultimately improve outcomes for children with ADHD. The automated algorithms and decision rules the investigators have developed for creating and monitoring the behavioral tools ensure that behavioral treatments like daily report cards and token economies are delivered in a manner that is consistent with the evidence-base. The investigators are conducting a cluster randomized controlled trial in community pediatric settings to test whether integration of the behavioral tools into the myADHDportal.com software (1) increases rates of behavioral treatment; (2) facilitates better integrity of behavioral interventions when implemented; (3) improves functional impairment in children with ADHD; and (4) generates higher satisfaction with ADHD care. By continuing to expand the functionality of the myADHDportal.com software, the investigators are increasing patients' access to evidence-based care. This is especially critical for rural and underserved communities who have no or limited access to evidence-based mental health services. Moreover, by putting these behavioral tools in the hands of parents, teachers, and pediatricians, the investigators are making it more likely that children will receive a high quality of care that includes both medication management and behavioral strategies, thereby improving the overall treatment outcomes of children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* child in grades K-5
* child has been diagnosed with ADHD by pediatrician or other mental health professional
* child's ADHD care is currently being managed by pediatrician
* if child is being prescribed ADHD medication, is currently on a stable dosage of medication
* child is experiencing impairment at school as evidenced by a rating of 3 or higher on parent- or teacher-ratings of "academic progress" or "problems in classroom" and on the Impairment Rating Scale.

Exclusion Criteria:

* parent does not have access to a computer or smartphone

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mehealth Portal With Integrated Behavioral Tools: Patients in this arm will have access to online behavioral interventions such as daily report cards online integrated within mehealth for attention deficit hyperactivity disorder (ADHD) software that allows parents and teachers to set up and deliver behavioral interventions such as daily report card systems and home-based program such as star charts.
- Mehealth Portal With no Integrated Behavioral Tools: Patients in this arm will wait one year before getting access to the behavioral intervention features.
Period: Overall Study
Arm/Group | Mehealth Portal With Integrated Behavioral Tools | Mehealth Portal With no Integrated Behavioral Tools
Started | 85 | 84
6-month Timepoint | 63 | 79
12-month Timepoint | 53 | 75
Completed | 53 | 75
Not Completed | 32 | 9
Not completed — Lost to Follow-up | 16 | 8
Not completed — Withdrawal by Subject | 16 | 1

BASELINE CHARACTERISTICS:
Groups:
- Mehealth Portal With Integrated Behavioral Tools: Patients in this arm will have access to online behavioral interventions such as daily report cards online integrated within mehealth for ADHD software that allows parents and teachers to set up and deliver behavioral interventions such as daily report card systems and home-based program such as star charts
- Total: Total of all reporting groups
Arm/Group | Mehealth Portal With Integrated Behavioral Tools | Mehealth Portal With no Integrated Behavioral Tools | Total
Number analyzed (Participants) | 85 | 84 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 85 | 84 | 169
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.23 (1.67) | 8.95 (1.71) | 9.09 (1.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 61 | 55 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 81 | 164
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 71 | 69 | 140
  More than one race | 5 | 8 | 13
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 85 | 84 | 169
Parent-report of child receiving behavioral treatment at home or school [Number; unit: participants] — Collected via parent-report using Services Use in Children and Adolescents Parent Interview
  participants | 70 | 66 | 136
Parent rating of School Performance on Impairment Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Parent rating of child's impairment on School Performance on the Impairment Rating Scale. Items rated on a Likert scale ranging from 0 (no impairment) to 6 (extreme impairment).
  units on a scale | 3.27 (1.85) | 3.64 (1.73) | 3.46 (.179)
Teacher rating of Academic Performance on Impairment Rating Scale [Mean (Standard Deviation); unit: units on a scale] | 3.15 (1.79) | 3.45 (1.69) | 3.30 (1.79)
Teacher rating of Classroom Performance on Impairment Rating Scale [Mean (Standard Deviation); unit: units on a scale] | 2.66 (1.76) | 2.55 (1.95) | 2.60 (1.85)

OUTCOME MEASURES:

1. Primary Outcome: Rates of Behavioral Treatment
Description: Parent-report of implementation of behavioral interventions on the Services Use in Children and Adolescents Parent Interview
Time Frame: 12 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Mehealth Portal With Integrated Behavioral Tools | Mehealth Portal With no Integrated Behavioral Tools
Number analyzed (Participants) | 85 | 84
Participants | 44 | 64
Statistical Analysis 1: Comparison: Mehealth Portal With Integrated Behavioral Tools vs Mehealth Portal With no Integrated Behavioral Tools; Test type: Superiority; p = .535, Chi-squared; Odds Ratio (OR) = .384

2. Secondary Outcome: Parent Rating of School Performance on Impairment Rating Scale
Description: Parent rating of child's impairment on School Performance on the Impairment Rating Scale. Items rated on a Likert scale ranging from 0 (no impairment) to 6 (extreme impairment).
Time Frame: 6 months after randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mehealth Portal With Integrated Behavioral Tools | Mehealth Portal With no Integrated Behavioral Tools
Number analyzed (Participants) | 85 | 84
units on a scale | 3.14 (1.65) | 3.50 (1.48)
Statistical Analysis 1: Comparison: Mehealth Portal With Integrated Behavioral Tools vs Mehealth Portal With no Integrated Behavioral Tools; Test type: Superiority; p = .829, ANOVA; Slope = .018, Standard Error of Mean .081

3. Secondary Outcome: Teacher Rating of Academic Performance on Impairment Rating Scale
Description: Teacher rating of child's impairment on Academic Performance on the Impairment Rating Scale. Items rated on a Likert scale ranging from 0 (no impairment) to 6 (extreme impairment).
Time Frame: 6 months after randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mehealth Portal With Integrated Behavioral Tools | Mehealth Portal With no Integrated Behavioral Tools
Number analyzed (Participants) | 62 | 62
units on a scale | 2.87 (1.95) | 3.38 (1.69)
Statistical Analysis 1: Comparison: Mehealth Portal With Integrated Behavioral Tools vs Mehealth Portal With no Integrated Behavioral Tools; Test type: Superiority; p = .357, ANOVA; Slope = -.105, Standard Error of Mean .093

4. Secondary Outcome: Teacher Rating of Classroom Performance on Impairment Rating Scale
Description: Teacher rating of child's impairment on Classroom Performance on the Impairment Rating Scale. Items rated on a Likert scale ranging from 0 (no impairment) to 6 (extreme impairment).
Time Frame: 6 months after randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mehealth Portal With Integrated Behavioral Tools | Mehealth Portal With no Integrated Behavioral Tools
Number analyzed (Participants) | 62 | 62
units on a scale | 2.27 (1.82) | 2.21 (1.78)
Statistical Analysis 1: Comparison: Mehealth Portal With Integrated Behavioral Tools vs Mehealth Portal With no Integrated Behavioral Tools; Test type: Superiority; p = .782, ANOVA; Slope = -.035, Standard Error of Mean .126

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Mehealth Portal With Integrated Behavioral Tools | Mehealth Portal With no Integrated Behavioral Tools
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/84
Other Adverse Events (participants affected / at risk) | 0/85 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03628781/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT03628781/ICF_001.pdf